CLINICAL TRIAL: NCT04043052
Title: MObile Technologies In the preVention of POSt-stroke DEPression
Brief Title: Mobile Technologies and Post-stroke Depression
Acronym: MOTIV-POSDEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2017/49
Record Dates: First submitted 2019-07-25; First posted 2019-08-02 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Depression
Keywords: Stroke; e-health; Depression; Anxiety; Prevention
MeSH Terms: conditions — Stroke; Depression; Anxiety Disorders | interventions — Ecological Momentary Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual (TAU) (Active Comparator): Evaluation of depression and anxiety disorders at 3 and 6 months post-stroke using psychological and functional examination
  Interventions: Other: Psychological evaluation; Other: Functional evaluation; Biological: Biological assessment
- EMA intervention assocuated to Treatment As Usual (EMA-TAU) (Experimental): Evaluation of depression and anxiety disorders at 3 and 6 months post-stroke using psychological and functional examination in addition with Ecological Momentary Assessment (EMA) evaluation.
  Interventions: Other: Psychological evaluation; Other: Functional evaluation; Biological: Biological assessment; Other: Ecological Momentary Assessment

INTERVENTIONS:
Other: Psychological evaluation — Psychological evaluation including: MINI (current diagnosis) ; HDRS ; MDQ ; GAD-7 ; PC-PTSD-5 ; Quality of Sleep (item 6 of the Pittsburgh Sleep Quality Index) ; CES-D ; BAI ; RRS-short form ; IES-R ; mYFAS2.0;
Other: Functional evaluation — Functional evaluation including : EQ5-D ; MFI ; LUNS ; SSQ ; Physical activity (IPAQ)
Biological: Biological assessment — Biological assessment : White and red blood cells count ; platelets count ; Haemoglobin ; CRPus ; Glycaemia ; Plasmatic HbA1c ; Plasmatic LDLc ; HDLc and triglyceride ; Creatinin clearance, Transaminases.
Other: Ecological Momentary Assessment — During 3 months after inclusion, a 3 to 5 minutes daily interview will administer questions concerning mood symptoms, activities, stress experience, substance use, social relationships and medication intake, activities, social interaction, environmental conditions, experience of depressed mood, anhedonia, changes in weight, appetite, sleep, fatigue, feelings of worthlessness or inappropriate guilt, concentration or decision-making difficulty
  Arms: EMA intervention assocuated to Treatment As Usual (EMA-TAU)

SUMMARY:
The recent development of acute phase treatments has dramatically improved stroke functional outcome but post-stroke neuropsychiatric disorders, notably post-stroke depression, continue to contribute to the heavy burden of stroke. While these conditions affect about 25% of stroke patients at 3 months, they are under-reported spontaneously by patients and are under-evaluated and treated by clinicians. Other than stroke severity and psychiatric history, risk factors for post-stroke depression remain a matter of debate, thus preventing identification of high-risk patients. Moreover, to date, neither pharmacological nor nonpharmacological treatments have demonstrated a significant benefit in the prevention of this disorder, thereby also impeding the development of early treatment strategies. Yet,the early management of post-stroke depression is critical given its negative influence on long-term functional outcomes, medication adherence, efficient use of rehabilitation services and the risk of stroke recurrence or vascular events. There is a pressing need to develop new tools allowing for the early detection of post-stroke neuropsychiatric complications for each individual patient. The rapid expansion of ambulatory monitoring techniques, such as Ecological Momentary Assessment (EMA), allows daily evaluations of mood symptoms in real time and in the natural contexts of daily life. The investigators have previously validated the feasibility and validity of EMA to assess daily life emotional symptoms after stroke, demonstrating its utility to investigate their evolution during the 3 months following stroke and to identify early predictors of post-stroke depression such as stress reactivity and social support, suggesting that EMA could be used in the early personalized care management of these neuropsychiatric complications. Recently, preliminary data have also emphasized the potential of EMA interventions to improve the outcome of psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Male or Female.
* Recent (≤ 15 days) clinically-symptomatic ischemic or hemorrhagic stroke documented through brain imaging (CT or MRI) or a Transient Ischemic Attack with an ABCD2 score ≥ 4.
* Patient discharged to home after hospitalization in the stroke unit.
* No severe neurological handicap: modified Rankin scale ≤ 3 at inclusion.
* No severe cognitive impairment or dementia: MoCA ≥ 16 at inclusion.
* Written informed consent by the patient.
* Covered by French Social Insurance

Exclusion Criteria:

* Transient Non Cerebrovascular Event.
* Subarachnoid hemorrhage.
* Dementia syndrome or other neurologic disorder and/or severe aphasia (NIHSS item 9 ≥ 2) interfering with the completion of evaluations and the utilization of EMA.
* Severe visual impairment interfering with the utilization of EMA.
* Severely impaired physical and/or mental health that, according to the investigator, may affect the participant's compliance with the study
* Patients with a severe substance use disorder (DSM-5 criteria)
* Patients under antidepressant and/or anxiolytic and/or neuroleptic and/or mood stabilizer treatment during the month preceding inclusion
* Participation in another protocol modifying the patient's follow-up status.
* Pregnancy or breastfeeding
* Inability to read French or to use a smartphone
* Individuals under legal protection or unable to express personnally their consent
* Individuals living in an area without 3G/4G internet coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2025-03-23 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale score (HDRS) | Day 0
  Semi-structured interview questionnaire designed to be used by a health care professional to investigate depressive symptomatology. 17 items are used to provide a score.
Hamilton Depression Rating Scale score (HDRS) | 3 months
  Semi-structured interview questionnaire designed to be used by a health care professional to investigate depressive symptomatology. 17 items are used to provide a score.
Hamilton Depression Rating Scale score (HDRS) | 6 months
  Semi-structured interview questionnaire designed to be used by a health care professional to investigate depressive symptomatology. 17 items are used to provide a score.

SECONDARY OUTCOMES:
Mini International Neuropsychiatric Interview (MINI) | Day 0
Mini International Neuropsychiatric Interview (MINI) | 3 months
Mini International Neuropsychiatric Interview (MINI) | 6 months
Mood Disorder Questionnaire (MDQ) | 3 months
  13 questions on mood symptoms and 2 additional questions on the co-occurrence and psychosocial impact of these symptoms. This questionnaire assesses the probability of an existing bipolar disorder. A positive screen include : a) answering 'Yes' to at least 7 of 13 questions, and b) reporting that several of these symptoms have been experienced during the same period of time, and c) reporting that psychosocial impairment has been caused by these symptoms.
Mood Disorder Questionnaire (MDQ) | 6 months
  13 questions on mood symptoms and 2 additional questions on the co-occurrence and psychosocial impact of these symptoms. This questionnaire assesses the probability of an existing bipolar disorder. A positive screen include : a) answering 'Yes' to at least 7 of 13 questions, and b) reporting that several of these symptoms have been experienced during the same period of time, and c) reporting that psychosocial impairment has been caused by these symptoms.
Generalized Anxiety Disorder-7 scale (GAD-7) | 3 months
  7 items that assess GAD symptoms experienced over the past two weeks. Patients are asked the frequency of these symptoms using a 4-point scale, ranging from 0 (Not at all) to 3 (Nearly every day). A cutoff score of greater than 10 is commonly used to identify cases of GAD.
Generalized Anxiety Disorder-7 scale (GAD-7) | 6 months
  7 items that assess GAD symptoms experienced over the past two weeks. Patients are asked the frequency of these symptoms using a 4-point scale, ranging from 0 (Not at all) to 3 (Nearly every day). A cutoff score of greater than 10 is commonly used to identify cases of GAD.
Primary Care PTSD Screen for DSM-5 (PC-PTSD-5) | 3 months
  5-item screen designed to identify individuals with probable PTSD. It begins with an item designed to assess whether the respondent has had any exposure to traumatic events. If a respondent denies exposure, the scale is completed with a score of 0. If the respondent indicates a trauma history, he/she has additional Yes/No questions about how the traumatic event has affected him/her over the past month. If the total score is 3 or more, the screen indicates probable PTSD.
Primary Care PTSD Screen for DSM-5 (PC-PTSD-5) | 6 months
  5-item screen designed to identify individuals with probable PTSD. It begins with an item designed to assess whether the respondent has had any exposure to traumatic events. If a respondent denies exposure, the scale is completed with a score of 0. If the respondent indicates a trauma history, he/she has additional Yes/No questions about how the traumatic event has affected him/her over the past month. If the total score is 3 or more, the screen indicates probable PTSD.
Center of Epidemiological Studies-Depression Scale (CES-D) | 3 months
  20-item. It measures symptoms of depression in nine different groups as defined by the DSM-5: Sadness (Dysphoria, 3 items), Loss of Interest (Anhedonia, 2 items), Appetite (2 items), Sleep (3 items), Thinking (Concentration, 2 items), Guilt or Worthlessness (2 items), Fatigue (2 items), Agitation (2 items), Suicidal ideation (2 items).
Center of Epidemiological Studies-Depression Scale (CES-D) | 6 months
  20-item. It measures symptoms of depression in nine different groups as defined by the DSM-5: Sadness (Dysphoria, 3 items), Loss of Interest (Anhedonia, 2 items), Appetite (2 items), Sleep (3 items), Thinking (Concentration, 2 items), Guilt or Worthlessness (2 items), Fatigue (2 items), Agitation (2 items), Suicidal ideation (2 items).
Beck Anxiety Inventory (BAI) | 3 months
  The Beck Anxiety Inventory (BAI) assesses the severity of patient anxiety during the past week. Though anxiety can be thought of as having several components, including cognitive, somatic, affective, and behavioral components included only two components in the BAI's original version: cognitive and somatic symptoms, with the cognitive subscale providing a measure of fearful thoughts and impaired cognitive functioning whereas the somatic subscale measures the symptoms of physiological arousal. Care was taken during scale construction to eliminate items that would be confounded with depression items. Patients respond to the frequence of 21 symptoms using a scale from 0 (Never) to 3 (Frequently, Almost every day).
Beck Anxiety Inventory (BAI) | 6 months
  The Beck Anxiety Inventory (BAI) assesses the severity of patient anxiety during the past week. Though anxiety can be thought of as having several components, including cognitive, somatic, affective, and behavioral components included only two components in the BAI's original version: cognitive and somatic symptoms, with the cognitive subscale providing a measure of fearful thoughts and impaired cognitive functioning whereas the somatic subscale measures the symptoms of physiological arousal. Care was taken during scale construction to eliminate items that would be confounded with depression items. Patients respond to the frequence of 21 symptoms using a scale from 0 (Never) to 3 (Frequently, Almost every day).
Ruminative Response Scale-short form (RRS-short form) | 3 months
  Ruminative Response Scale-short form (RRS-short form) is one of the most widely used self-reported measures of rumination, comprising 9 items and describing the factors of brooding (5 items) and reflection (5 items). For each item, patients indicate the frequency of each event on a 4-point scale ranging from 1 ("almost never") to 4 ("almost always").
Ruminative Response Scale-short form (RRS-short form) | 6 months
  Ruminative Response Scale-short form (RRS-short form) is one of the most widely used self-reported measures of rumination, comprising 9 items and describing the factors of brooding (5 items) and reflection (5 items). For each item, patients indicate the frequency of each event on a 4-point scale ranging from 1 ("almost never") to 4 ("almost always").
Multidimensional Fatigue Inventory (MFI) | 3 months
  The MFI contains 20 items classified into four dimensions: general fatigue, mental fatigue, reduced activities and motivation. The statements are rated on a 5-point Likert scale (from "Yes, that is true" to "No, that is not true") representing the patient's current feeling. Low MFI scores reflect a higher degree of fatigue.
Multidimensional Fatigue Inventory (MFI) | 6 months
  The MFI contains 20 items classified into four dimensions: general fatigue, mental fatigue, reduced activities and motivation. The statements are rated on a 5-point Likert scale (from "Yes, that is true" to "No, that is not true") representing the patient's current feeling. Low MFI scores reflect a higher degree of fatigue.
EuroQoL 5-Dimensions Questionnaire (EQ-5D) | 3 months
  The EuroQoL 5-Dimensions Questionnaire (EQ-5D) is a standardized instrument for use as a measure of health outcome in stroke and was designed for self-completion by respondents. The 5 items of the questionnaire provide a simple descriptive profile and a single index value for health status. The EQ-Index has shown reasonable validity and acceptable responsiveness for detecting the health-related quality of life in stroke patients.
EuroQoL 5-Dimensions Questionnaire (EQ-5D) | 6 months
  The EuroQoL 5-Dimensions Questionnaire (EQ-5D) is a standardized instrument for use as a measure of health outcome in stroke and was designed for self-completion by respondents. The 5 items of the questionnaire provide a simple descriptive profile and a single index value for health status. The EQ-Index has shown reasonable validity and acceptable responsiveness for detecting the health-related quality of life in stroke patients.
Long-term Unmet Needs after Stroke (LUNS) | 3 months
  The Long-term Unmet Needs after Stroke (LUNS) includes 22 items that have each been worded to ask whether the respondent has a need and whether the need is met, and the potential complexity of "double-barrelled" questions was managed by providing Yes or No response modalities, with instructions to tick 'No' if there is no need or if the need has been met. Participants are also asked to indicate what level of help (from care givers/friends) they have received in completing the questionnaires, if any.
Long-term Unmet Needs after Stroke (LUNS) | 6 months
  The Long-term Unmet Needs after Stroke (LUNS) includes 22 items that have each been worded to ask whether the respondent has a need and whether the need is met, and the potential complexity of "double-barrelled" questions was managed by providing Yes or No response modalities, with instructions to tick 'No' if there is no need or if the need has been met. Participants are also asked to indicate what level of help (from care givers/friends) they have received in completing the questionnaires, if any.
Short version of Sarason's Social Support Questionnaire (6 items SSQ) | 3 months
  Used to measure two dimensions of social support : satisfaction and availability perceptions of social support and satisfaction with that social support. Each item is a question that solicits a two-part answer: Part 1 asks participants to list all the people that fit the description of the question, and Part 2 asks participants to indicate how satisfied they are in general with these people using a 6-point Licket scale (from 1. Very unsatisfied to 6. Extremely satisfied).
Short version of Sarason's Social Support Questionnaire (6 items SSQ) | 6 months
  Used to measure two dimensions of social support : satisfaction and availability perceptions of social support and satisfaction with that social support. Each item is a question that solicits a two-part answer: Part 1 asks participants to list all the people that fit the description of the question, and Part 2 asks participants to indicate how satisfied they are in general with these people using a 6-point Licket scale (from 1. Very unsatisfied to 6. Extremely satisfied).
International Physical Activity Questionnaire (7 items IPAQ) | Day 0
  The International Physical Activity Questionnaire (7 items IPAQ) assesses physical activity undertaken across a comprehensive set of domains including: a. leisure time physical activity, b. domestic and gardening activities, c. work related physical activity, d. transport-related physical activity. The IPAQ short form asks about three specific types of activity undertaken in these four domains : walking, moderate-intensity activities and vigorous-intensity activities. Computation of the total score for the short form requires summation of the duration (in minutes) and frequency (days) of walking, moderate-intensity and vigorous-intensity activities.
International Physical Activity Questionnaire (7 items IPAQ) | 3 months
  The International Physical Activity Questionnaire (7 items IPAQ) assesses physical activity undertaken across a comprehensive set of domains including: a. leisure time physical activity, b. domestic and gardening activities, c. work related physical activity, d. transport-related physical activity. The IPAQ short form asks about three specific types of activity undertaken in these four domains : walking, moderate-intensity activities and vigorous-intensity activities. Computation of the total score for the short form requires summation of the duration (in minutes) and frequency (days) of walking, moderate-intensity and vigorous-intensity activities.
International Physical Activity Questionnaire (7 items IPAQ) | 6 months
  The International Physical Activity Questionnaire (7 items IPAQ) assesses physical activity undertaken across a comprehensive set of domains including: a. leisure time physical activity, b. domestic and gardening activities, c. work related physical activity, d. transport-related physical activity. The IPAQ short form asks about three specific types of activity undertaken in these four domains : walking, moderate-intensity activities and vigorous-intensity activities. Computation of the total score for the short form requires summation of the duration (in minutes) and frequency (days) of walking, moderate-intensity and vigorous-intensity activities.
Percentage of stroke risk | Day 0
  The Riskometer application will be used to measure the stroke risk based on recorded parameters. The Stroke Riskometer app assesses the possibility of suffering a stroke using a number of health and lifestyle factors including age, sex, ethnic origin, blood pressure, atrial fibrillation, left ventricular hypertrophy, anti-hypertension, tobacco, cardiovascular history, weight / height ratio, cholesterol level, diabetes, alcohol, stress, cognitive decline, family and personal history of stroke and TIA, history of head trauma and myocardial infarction
Percentage of stroke risk | 3 months
  The Riskometer application will be used to measure the stroke risk based on recorded parameters. The Stroke Riskometer app assesses the possibility of suffering a stroke using a number of health and lifestyle factors including age, sex, ethnic origin, blood pressure, atrial fibrillation, left ventricular hypertrophy, anti-hypertension, tobacco, cardiovascular history, weight / height ratio, cholesterol level, diabetes, alcohol, stress, cognitive decline, family and personal history of stroke and TIA, history of head trauma and myocardial infarction
Percentage of stroke risk | 6 months
  The Riskometer application will be used to measure the stroke risk based on recorded parameters. The Stroke Riskometer app assesses the possibility of suffering a stroke using a number of health and lifestyle factors including age, sex, ethnic origin, blood pressure, atrial fibrillation, left ventricular hypertrophy, anti-hypertension, tobacco, cardiovascular history, weight / height ratio, cholesterol level, diabetes, alcohol, stress, cognitive decline, family and personal history of stroke and TIA, history of head trauma and myocardial infarction
Recurrent stroke | 3 months
  Recurrent stroke or TIA post-stroke defined by standard clinico-radiological criteria
Recurrent stroke | 6 months
  Recurrent stroke or TIA post-stroke defined by standard clinico-radiological criteria
Cardiovascular events post-stroke | 3 months
  Cardiovascular events post-stroke defined by standard clinical criteria
Cardiovascular events post-stroke | 6 months
  Cardiovascular events post-stroke defined by standard clinical criteria
Intensity of post-stroke pain | Day 0
  Intensity of post-stroke pain using a visual analog scale
Intensity of post-stroke pain | 3 months
  Intensity of post-stroke pain using a visual analog scale
Intensity of post-stroke pain | 6 months
  Intensity of post-stroke pain using a visual analog scale
Pittsburgh Sleep Quality Index | Visit 1 ; 3 months ; 6 months
  Quality of sleep using the item 6 of the Pittsburgh Sleep Quality Index
Blood pressure | Visit 1 ; 3 months ; 6 months
  Blood pressure
HbA1c measure | 3 months ; 6 months
  Glycaemic control using the HbA1c measure
LDLc plasmatic measure | 3 months ; 6 months
  Lipidic control using the LDLc plasmatic measure
CRPus plasmatic measure | 3 months ; 6 months
  Systemic inflammation will be evaluated using CRPus plasmatic measure
Smoking Index (HSI) | 3 months ; 6 months
  Tobacco use will be evaluated using the Heaviness of Smoking Index (HSI)

CONTACTS AND LOCATIONS:
Overall Officials: Igor SIBON, Principal Investigator — University Hospital, Bordeaux
Locations (5):
- France (5):
  - CHU de Bordeaux, Bordeaux
  - CHRU de Brest, Brest
  - CHU Dijon Bourgogne, Dijon
  - CHU de Montpellier, Montpellier
  - Assistance Publique Hopitaux de Paris - Groupe Hospitalier Paris Saint Joseph, Paris

IPD SHARING:
Plan to Share IPD: No